CLINICAL TRIAL: NCT06798259
Title: Autonomic Dysfunction in Patients With Migraine: Cardiovascular and Neurophysiology Assessment
Status: Active, not recruiting | Type: Observational
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Donia Adel Abd-ElSadek, Assistant teacher of anesthesiology ,pain management and surgical ICU departement, Beni-Suef University
Other Study IDs: FMBSUREC/01102024/Abd-Elsadek
Record Dates: First submitted 2025-01-07; First posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Migraine Headache
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Autonomic dysfunction in patients with migraine: cardiovascular and neurophysiology assessment.

DETAILED DESCRIPTION:
assessment if Autonomic dysfunction in patients with migraine by using cardiovascular assessment by HOTLER MONITORING and table tilt test and neurophysiology assessment by sympathetic skin response

ELIGIBILITY:
Inclusion Criteria:

* 1.fulfilling ICHD-3 criteria for migraine 2. migraine for at least 3 months.

Exclusion Criteria:

brain imaging showing structural brain lesions. .medications that could impact autonomic function such as tricyclic antidepressants, anticholinergics, or opioids.

* Patients with concomitant medical illness causing autonomic dysfunction such as: diabetes, cardiovascular, demyelinating or degenerative neurological disorders.
* Contraindications for performing the tilt test
* Pregnant patients.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: . The patients will be recruited from the Neurology clinic, Beni Suef University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 116 (Estimated)
Dates: Start 2025-01-07 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Autonomic dysfunction in patients with migraine | baseline
  assessment of autonomic dysfunction using Composite autonomic system Score 31

SECONDARY OUTCOMES:
Cardiovascular assessment | 24 hours
  Cardiovascular is done using Holter monitoring and table tilt est

CONTACTS AND LOCATIONS:
Locations (1):
- Benisuef university hospital, Benisuef, Benisuef, Egypt